CLINICAL TRIAL: NCT07369284
Title: Efficacy of Melatonin in Addition to Standard Care in Glycemic Control of Patients With Gestational Diabetes Mellitus: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Melatonin for Glycemic Control in Gestational Diabetes Mellitus
Acronym: MELODY
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Collaborators: West China Second University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-260
Record Dates: First submitted 2026-01-05; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes; Melatonin; Fasting plasma glucose
MeSH Terms: conditions — Diabetes, Gestational | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): 1. Melatonin tablets will be administered orally 0.5 to 1 hour before sleep and at least 2 hours after the last meal.
  2. Participants will take 5 mg melatonin every night during the first week of intervention after randomization, followed by 10 mg melatonin every night from the second week until delivery.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): 1. Identical placebo tablets in terms of packaging, appearance, smell and taste will be administered orally 0.5 to 1 hour before sleep and at least 2 hours after the last meal.
  2. Participants will take identical placebo tablets after randomization until delivery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — 1. Melatonin tablets will be administered orally 0.5 to 1 hour before sleep and at least 2 hours after the last meal.
  2. Participants will take 5 mg melatonin every night during the first week of intervention after randomization, followed by 10 mg melatonin every night from the second week until delivery.
  Arms: Melatonin
Other: Placebo — 1. Identical placebo tablets in terms of packaging, appearance, smell and taste will be administered orally 0.5 to 1 hour before sleep and at least 2 hours after the last meal.
  2. Participants will take identical placebo tablets after randomization until delivery.
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to evaluate whether melatonin supplementation improves glycemic control in pregnant women diagnosed with gestational diabetes mellitus (GDM).

The main question it aims to answer is:

Does melatonin supplementation help with glycemic control, especially in lowering fasting plasma glucose level?

Researchers will compare melatonin to a placebo (a look-alike substance that contains no melatonin) to see if melatonin works to improve glycemic control.

Participants will:

1. Take melatonin or a placebo every day after randomization until delivery
2. Visit the antenatal clinic once every 1 to 2 weeks for follow-ups

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45 years
* Singleton pregnancy
* A diagnosis of GDM from a 75-g OGTT during 24 to 28 gestational weeks, according to the IADPSG criteria, with at least fasting plasma glucose (FPG) ≥ 5.1 mmol/L
* Intending to receive obstetric care and deliver in the study center
* Willing and able to provide written informed consent and follow the study procedure

Exclusion Criteria:

* Use of melatonin 1 month before pregnancy or/and during pregnancy
* Night shift work or exposed to jetlag on a regular basis during pregnancy
* Contraindications to melatonin use, including hypersensitive or allergic to melatonin
* Use of antidepressive or antipsychotic medications which can interfere with melatonin metabolism and/or elimination, such as fluvoxamine, 5- or 8-methoxypsoralen, cimetidine, quinolones, and other CYP1A2 inhibitors; carbamazepine, rifampicin, and other CYP1A2 inducers; and zaleplon, zolpidem, zopiclone, and other non-benzodiazepine hypnotics
* Pre-pregnancy diabetes, including patients diagnosed with diabetes before conception, fasting plasma glucose ≥ 7.0 mmol/L or HbA1c ≥ 6.5% in the first trimester, typical hyperglycemic symptoms or hyperglycemic crisis with random blood glucose ≥ 11.1 mmol/L
* Other major diseases before gestation, e.g. hypertensive disorders, rheumatology or malignant diseases, infected with hepatitis B or hepatitis C, chronic diseases leading to impaired heart, liver, or renal function
* Major fetal anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in fasting plasma glucose (FPG) from baseline to 36 to 38 gestational weeks | Baseline (24 to 28 gestational weeks), and 36 to 38 gestational weeks
  The primary outcome is defined as the change in FPG levels from baseline, measured at the time of OGTT performed between 24 and 28 gestational weeks, to follow-up assessment at 36 to 38 gestational weeks. For participants who deliver before 36 gestational weeks, the last available FPG measurement obtained will be used.

SECONDARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) from baseline to 36 to 38 gestational weeks | Baseline and 36 to 38 gestational weeks
  This outcome is defined as change in HbA1c levels from baseline, measured at the time of OGTT performed between 24 and 28 gestational weeks, to follow-up assessment at 36 to 38 gestational weeks.
Initiation of insulin therapy | From baseline until delivery
  This outcome is defined as the proportion of participants requiring initiation of insulin therapy.
Change in mean glucose levels assessed by continuous glucose monitoring (CGM) | Baseline and 36 to 38 gestational weeks
  This outcome is defined as the change in mean glucose levels measured by CGM at baseline and before delivery.
Gestational weight gain in late pregnancy | From baseline until delivery
  This outcome is defined as total gestational weight gain and the rate of weight gain from baseline to the last assessment prior to delivery.
Incidence of intervention-related adverse events | From initiation of the intervention until 6 weeks postpartum
  This outcome is defined as the proportion of participants reporting adverse events potentially related to study intervention, including but not limited to dizziness, hypersomnia, nausea, vomiting and hypoglycemia. Adverse events will be collected from participants' medication diaries and systematically assessed through participant self-report at each antenatal clinic visit.
Impact of melatonin on fetal growth | From baseline until delivery
  The antenatal use of melatonin on estimated fetal growth (grams) will be assessed using ultrasound biometry parameters performed every two to four weeks following trial recruitment until birth.
Percentage of time in range, time above range, and time below range measured by CGM | Baseline and 36 to 38 gestational weeks
  This outcome is defined as percentages of time in range, time above range, and time below range measured by CGM at baseline and before delivery.

OTHER OUTCOMES:
Pregnancy complications | From baseline until the end of follow-up at 6 weeks postpartum
  This outcome is defined as a series of pregnancy complications including but not limited to gestational hypertensive disorders and intrahepatic cholestasis of pregnancy.
Perinatal outcomes | From baseline until the end of follow-up at 6 weeks postpartum
  This outcome is defined as a series of perinatal outcomes including but not limited to the percentages of macrosomia, large for gestational age, small for gestational age, neonatal hypoglycemia, birth trauma, cesarean section, postpartum hemorrhage, placenta abruption, and spontaneous premature rupture of membranes.

IPD SHARING:
Plan to Share IPD: No